CLINICAL TRIAL: NCT02447237
Title: Randomized Controlled Trial About the Effect of Liquid Compared to Solid Food on the Intake of Energy and Protein in Patients With Leukemia, Lymphoma or Other Malignant Hematologic Disease
Brief Title: Randomized Trial:the Effect of Liquid Food on the Intake of Energy and Protein in Malignant Hematologic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Rikardt Andersen (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor at Department of Nutrition, Exercise and Sports, University of Copenhagen, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-4-2014-113
Record Dates: First submitted 2015-03-25; First posted 2015-05-18 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Hematological Disease; Delayed Gastric Emptying; Malignant Disease
Keywords: liquid diet; solid diet
MeSH Terms: conditions — Hematologic Diseases; Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- liquid food (Experimental): dietary counselling in fulfilling need of protein and energy through liquid food
  Interventions: Other: dietary counselling
- solid food (Other): dietary counselling in fulfilling need of protein and energy through solid food
  Interventions: Other: dietary counselling

INTERVENTIONS:
Other: dietary counselling — the participants will receive dietary counselling in fulfilling their need of energy and protein according to the group they are randomized to (either solid or liquid food).

SUMMARY:
The study investigates the effect of liquid food on the intake of energy and protein compared to solid food. One group will receive dietary counselling in fulfilling their need for energy and protein from liquid food and the other group from solid food.

DETAILED DESCRIPTION:
The study investigates the effect of liquid food on the intake of energy and protein compared to solid food. One group will receive dietary counselling in fulfilling their need for energy and protein from liquid food and the other group from solid food. Both groups need to register their dietary intake in a period of 14 days and will be weighed three times during the intervention. At the end of the intervention they need to fill out a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* patients with leukemia, lymphoma or other malignant hematological disease
* adults
* be able to talk and understand danish
* be able to eat both solid and liquid food

Exclusion Criteria:

* not able to cooperate
* need for total tube or parenteral nutrition
* need for dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Intake of energy and protein | 14 days
  assessed by dietary records from both groups

SECONDARY OUTCOMES:
Weightloss change in percent from baseline | 14 days
  calculated by comparing baseline weight with the weight after 14 days
Amount of infections | 14 days
  infection, e.g. fever, diarrhoea will be assessed from the medical record
Need for tube feeding and parenteral nutrition | 14 days
  will be assessed from the medical record
patient satisfaction as well as perception of own nutritional status | 14 days
  will be assessed from a questionnaire filled out by the patient after completing the intervention
patients compliance of following the nutritional guidelines in the liquid group | 14 days
  calculating the amount of energy from liquid food compared to the total energy intake using the dietary records
Dose of cytostatics | 14 days
  will be assessed from the medical records
unplanned hospital stay | 14 days
  will be assessed from the medical record

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, Lektor, Study Director — Rigshospitalet, Denmark
Locations (1):
- Hematological clinic, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No